CLINICAL TRIAL: NCT03403634
Title: Phase 2a Study Evaluating a Chemokine-Modulatory Regimen in Patients With Colorectal Cancer Metastatic to the Liver
Brief Title: Celecoxib, Recombinant Interferon Alfa-2b, and Rintatolimod in Treating Patients With Colorectal Cancer Metastatic to the Liver
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 52917; NCI-2017-02471 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 52917 (Other: Roswell Park Cancer Institute); P01CA234212 (NIH)
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Metastatic Carcinoma in the Liver; Recurrent Colorectal Carcinoma; Stage IV Colorectal Cancer AJCC v7; Stage IVA Colorectal Cancer AJCC v7; Stage IVB Colorectal Cancer AJCC v7
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Celecoxib; Introns; Interferon alpha-2; poly(I).poly(c12,U)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (celecoxib, interferon alfa-2b, rintatolimod) (Experimental): Patients receive celecoxib orally PO BID, recombinant interferon alfa-2b IV QD over 20 minutes, and rintatolimod IV QD on days 1, 2, 3, 8, 9, 10, 15, 16 and 17 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Celecoxib; Other: Laboratory Biomarker Analysis; Biological: Recombinant Interferon Alfa-2b; Drug: Rintatolimod

INTERVENTIONS:
Drug: Celecoxib — Given PO
  Other Names: Benzenesulfonamide, 4-[5-(4-methylphenyl)-3-(trifluoromethyl)-1H-pyrazol-1-yl]-; Celebrex; SC-58635; YM 177
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Recombinant Interferon Alfa-2b — Given IV
  Other Names: Alfatronol; Glucoferon; Heberon Alfa; IFN alpha-2B; Interferon alfa 2b; Interferon Alfa-2B; Interferon Alpha-2b; Intron A; Sch 30500; Urifron; Viraferon
Drug: Rintatolimod — Given IV
  Other Names: Ampligen; Atvogen

SUMMARY:
This early phase IIA trial studies how well celecoxib, recombinant interferon alfa-2b, and rintatolimod work in treating patients with colorectal cancer that as spread to the liver. Celecoxib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Recombinant interferon alfa-2b is a substance that can improve the body's natural response and may interfere with the growth of tumor cells. Rintatolimod may stimulate the immune system. Giving celecoxib, recombinant interferon alfa-2b, and rintatolimod may work better at treating colorectal cancer that has spread to the liver.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the impact of a chemokine-modulatory regimen on the immune microenvironment of colorectal liver metastases, specifically the changes in the ratio between cytotoxic T-lymphocyte (CTL) marker (CD8a gene expression) to regulatory T cell (Treg) markers (FoxP3 gene expression).

SECONDARY OBJECTIVES:

I. Estimate the objective response rate of a chemokine-modulatory regimen in metastatic colorectal cancer (per Response Evaluation Criteria in Solid Tumors [RECIST] 1.1).

II. Examine the safety and tolerability profile of the combination of recombinant interferon alfa-2b (interferon alpha-2b), rintatolimod, and celecoxib when given as chemokine modulation to colorectal cancer patients prior to surgical resection using the Cancer Therapy Evaluation Program (CTEP) National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE version 4.0).

TERTIARY OBJECTIVES:

* Estimate the median progression free survival of a chemokine-modulatory regimen in metastatic colorectal cancer
* Estimate overall survival in participants with recurrent and/or metastatic unresectable colorectal cancer who received the chemokine-modulatory regimen
* Comparison (using RT-PCR, immunofluorescence [IF] and immunohistochemistry [IHC] on serial sections) of the metastatic tissue specimen with regard to total numbers of infiltrating T cells, their CD4/CD8 ratios, frequencies of FoxP3 cells, and the expression of chemokine receptors on CD4+ and CD8+ T cells (CXCR3, CCR5, CCR4, CCR6, and CXCR4)
* Evaluate the local expression of effector T cells (Teff)-attracting chemokines (CCR5, CXCL9, CXCL10 and CXCL11) and Treg-favoring chemokines (CCL22 and CXCL12) using IF and RT-PCR.

OUTLINE:

Patients receive celecoxib orally (PO) twice daily (BID), recombinant interferon alfa-2b intravenously (IV) over 20 minutes, and rintatolimod IV QD on days 1, 2,3,8,9,10,15,16 and 17 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent and/or metastatic unresectable colorectal cancer with hepatic metastases
* Hepatic metastases present which are amenable to biopsy
* Prior treatment with, contra-indication to or refusal of a fluoropyrimidine, irinotecan, oxaliplatin and an anti-EGFR targeted therapy (if RAS wild-type [wt]) as well as a PD-1 or PD-L1 targeted drug if MSI-H/dMMR
* No chemotherapy, radiotherapy, major surgery, or biologic therapy within 3 weeks of protocol treatment
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Have measurable disease per RECIST 1.1 criteria present
* Ability to swallow and retain oral medication
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Platelet >= 75,000/uL
* Hemoglobin >= 9 g/dL
* Hematocrit >= 27%
* Absolute neutrophil count (ANC) >= 1500/uL
* Creatinine < = institutional upper limit of normal (ULN) OR
* Creatinine clearance >= 50 mL/min for patients with creatinine levels greater than ULN
* Total bilirubin =< 1.5 X institutional ULN or for patients with known Gilbert's Syndrome total bilirubin <= 3 x ULN
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional ULN
* Plasma amylase =< 1.5 X institutional ULN
* Lipase =< 1.5 X institutional ULN
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Patients currently treated with systemic immunosuppressive agents, including steroids, are ineligible until 3 weeks after removal from immunosuppressive treatment
* Patients with active autoimmune disease, requiring ongoing immunosuppressive therapy or history of transplantation
* Patients who are pregnant or nursing; women of childbearing potential (WOCBP) will have to undergo a urine pregnancy test as part of screening
* Untreated central nervous system (CNS) metastases
* Cardiac risk factors including:

  * Patients experiencing cardiac event(s) (acute coronary syndrome, myocardial infarction, or ischemia) within 3 months of signing consent
  * Patients with a New York Heart Association classification of III or IV
* History of upper gastrointestinal ulceration, upper gastrointestinal bleeding, or upper gastrointestinal perforation within the past 3 years; patients with ulceration, bleeding or perforation in the lower bowel are not excluded
* Prior allergic reaction or hypersensitivity to celecoxib, or non-steroidal antiinflammatory drugs (NSAIDs) or any study agents which would prevent completion of protocol therapy
* Patients are ineligible if they plan on regular use of NSAIDs at any dose more than 2 times per week (on average) or aspirin at more than 325 mg at least three times per week, on average; low-dose aspirin not exceeding 100 mg/day is permitted; patients who agree to stop regular NSAIDs or higher dose aspirin are eligible and no wash out period is required
* Received an investigational agent within 30 days prior to enrollment
* Unwilling or unable to follow protocol requirements
* Patients with known serious mood disorders
* Any additional condition which in the investigator?s opinion deems the participant an unsuitable candidate to receive the study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2021-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarbajit Mukherjee, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Celecoxib, Interferon Alfa-2b, Rintatolimod)
Started | 19 (19 patients were accrued and completed consent.)
Treated | 15 (4 patients became ineligible prior to the start of treatment.)
Completed | 12
Not Completed | 7
Not completed — Disease progression | 3
Not completed — Did not meet eligibility criteria | 4

BASELINE CHARACTERISTICS:
Population: There were 19 patients accrued to the study; however, 4 never received any treatment and became ineligible.
Arm/Group | Treatment (Celecoxib, Interferon Alfa-2b, Rintatolimod)
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
Line of Treatment [Count of Participants; unit: Participants] — What line of treatment is the subject receiving 9i.e. number of prior lines + 1).
  Participants
    Third Line | 5
    Fourth Line | 6
    Fifth or More Line | 4
Clinical Stage [Count of Participants; unit: Participants] — Assessed by American Joint Committee on Cancer (AJCC) cancer staging system, 7th edition. Clinical Staging determines how much cancer there is based on the physical examination, imaging tests, and biopsies of affected areas.
  Stage I - lowest level of disease Stage IV - highest level of disease, with metastatic components
  Participants
    Stage I | 0
    Stage II | 0
    Stage III | 0
    Stage IV | 15
    Not Reported | 0
Location of Disease [Count of Participants; unit: Participants]
  Cecum | 1
  Colon, NOS | 7
  Rectum, NOS | 6
  Sigmoid Colon | 1
Prior Radiation [Count of Participants; unit: Participants] — Number of patients that received radiation as a prior therapy.
  Participants | 6
Prior Surgery [Count of Participants; unit: Participants] — Number of patients that had site specific surgery as part of a prior therapy.
  Participants | 10
RAS Type [Count of Participants; unit: Participants] — RAS mutation type was assessed using tumor tissue, and identified as either: KRAS mutation, NRAS mutation, or Wildtype.
  this was assessed as part of the inclusion criteria #3:
  "Prior treatment with, contra-indication to or refusal of a fluoropyrimidine, irinotecan, oxaliplatin and an anti-EGFR targeted therapy (if RAS wild type), as well as a PD-1 or PD-L1 targeted drug if MSI-H/dMMR."
  Participants
    KRAS | 5
    NRAS | 3
    Wild-type | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Tumor-infiltrating Lymphocytes (TILs) in the Colorectal Cancer Lesions
Description: The TILs will be summarized by time-point (pre-/post-treatment) using the mean, median, standard deviation; and graphically using dot-plots.
  The TIL of interest is CD8a expression, which is reported as the mean fold change from pre-treatment (i.e. post treatment / pre treatment).
Time Frame: Baseline up to 12 months
Population: 3 patients did not have post treatment biopsies, and were considered unevaluable for the primary endpoint.
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Treatment (Celecoxib, Interferon Alfa-2b, Rintatolimod)
Number analyzed (Participants) | 12
fold change | 7.25 (13.79)
Statistical Analysis 1: Comparison: Treatment (Celecoxib, Interferon Alfa-2b, Rintatolimod); Test type: Superiority; p = 0.046, t-test, 1 sided — significance level = 0.05; df = 11. one-sided as post treatment increases were of interest. the fold changes were log-transformed prior to inferences

2. Secondary Outcome: Number of Participants With Indicated Grade Adverse Event
Description: Safety profile will be characterized by type, frequency, severity, timing, seriousness and relationship to study treatment. The highest grade treatment related AE is provided (per Common Terminology Criteria for Adverse Events version 4.0).
Time Frame: Up to 12 months
Population: All patients that received study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Celecoxib, Interferon Alfa-2b, Rintatolimod)
Number analyzed (Participants) | 15
Participants
  No Treatment Related AE Reported | 1
  Grade I | 6
  Grade II | 7
  Grade III | 1
  Grade IV | 0
  Grade V | 0

3. Secondary Outcome: Objective Response Rate (ORR) Assessed by Response Evaluation Criteria in Solid Tumors Version (RECIST) 1.1
Description: Will be treated as binary data and summarized using frequencies and relative frequencies; with the ORR estimated using a 90% confidence interval obtained using Jeffrey's prior method.
Time Frame: Up to 12 months
Population: Evaluated in subjects evaluable for the primary end-point.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Celecoxib, Interferon Alfa-2b, Rintatolimod)
Number analyzed (Participants) | 12
Participants | 0

4. Other Pre Specified Outcome: Progression Free Survival
Description: Will be treated as bivariate time-to-event data and will be summarized using standard Kaplan-Meier methods.
Time Frame: From the start of treatment until disease progression (defined by RECIST 1.1) or last-follow-up, assessed up to 12 months
Population: Evaluated in subjects evaluable for the primary end-point.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Treatment (Celecoxib, Interferon Alfa-2b, Rintatolimod)
Number analyzed (Participants) | 12
Months | 1.5 [1.4 to 1.8]

5. Other Pre Specified Outcome: Overall Survival
Description: Will be treated as bivariate time-to-event data and will be summarized using standard Kaplan-Meier methods.
Time Frame: From the start of treatment until death due to any cause or last follow-up, assessed up to 12 months
Population: Evaluated in subjects evaluable for the primary end-point.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Treatment (Celecoxib, Interferon Alfa-2b, Rintatolimod)
Number analyzed (Participants) | 12
Months | 10.5 [2.2 to 15.2]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected up to 30 days after end of treatment, up to 1 year.
Arm/Group | Treatment (Celecoxib, Interferon Alfa-2b, Rintatolimod)
All-Cause Mortality (participants affected / at risk) | 8/15
Serious Adverse Events (participants affected / at risk) | 3/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Celecoxib, Interferon Alfa-2b, Rintatolimod) (N=15)
Hyperbilirubinemia (Hepatobiliary disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Neoplasm (NOS) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Celecoxib, Interferon Alfa-2b, Rintatolimod) (N=15)
Gastrointestinal disorders **Any AE - Maximum Grade Seen Diarrhoea (Gastrointestinal disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (2)
Asthenia (General disorders) | 1 (1)
Chills (General disorders) | 11 (11)
Fatigue (General disorders) | 11 (11)
Influenza like illness (General disorders) | 1 (1)
Pyrexia (Gastrointestinal disorders) | 5 (5)
Mucosal infection (Infections and infestations) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 1 (1)
Weight decreased (Investigations) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flush (Vascular disorders) | 6 (6)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/34/NCT03403634/Prot_SAP_000.pdf